CLINICAL TRIAL: NCT02040740
Title: Pubertal Assessment of Kidney-Bone Crosstalk
Brief Title: Mediators of Kidney-Bone Communication in Childhood
Acronym: PAKC
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Krista Casazza, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: PAKC
Record Dates: First submitted 2013-12-20; First posted 2014-01-20 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Fasting Blood Measures; Body Scans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma DNA collected to obtain ancestry informative markers and single nucleotide polymorphisms involved in mineral metabolism
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Healthy early pubertal boys

SUMMARY:
An identified hormone linking bone and kidney function is Fibroblast Growth Factor-23 (FGF23). Data on the variation of FGF23 levels for bone and mineral metabolism in children are scarce. Currently it is assumed that meeting mineral requirements for the skeleton serves the body's overall needs. However, it is not clear as to whether this is true, particularly with growth. The contribution of dietary factors directly linked with the bone/kidney axis through measurement of intake (via 24hr recall) and kidney nutrient clearance (via serum and urinary analysis) will be included in investigations. Findings will serve as a springboard for delineating more specific mechanisms by which these systems become disordered and are influenced by diet. It is expected that adequacy of nutrients known to have a central role in bone function will optimize the hormonal milieu through crosstalk with the kidney.

This effort will allow ongoing investigation in detecting and treating disturbances in mineral metabolism related to kidney disease, specifically in the pediatric population and broaden the understanding of kidney disease itself, as well as that of chronic diseases in which kidney health is of importance, such as diabetes and osteoporosis. Findings of this research may stress the importance of achieving dietary adequacy essential for establishing optimal body composition trajectories, particularly puberty.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ages 7-11y
* Tanner stage less than or equal to 3 according to the criteria of Marshall and Tanner

Exclusion Criteria:

* History of Cushing's Syndrome, hyperprolactinemia, congenital (non-classic) adrenal hyperplasia, type 1 or 2 diabetes, disturbances in glucose or lipid metabolism
* use of tobacco or consumption of alcohol; thyroid medication, diuretics, beta-blockers, or any medication that potentially could affect body composition, the lipid profile, insulin sensitivity, or blood pressure
* eating disorders, cancer, kidney disease, endocrinopathy, liver disease, heart disease, or thyroid disease.

Ages: 7 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy boys ages 7-11y
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Fibroblast Growth Factor 23 | 1 day
  Fasting plasma measure

CONTACTS AND LOCATIONS:
Overall Officials: Krista Casazza, PhD, RD, Principal Investigator — UAB, Nutrition Sciences; Orlando M Gutierrez, MD, Study Director — UAB, Department of Medicine; Lynae J Hanks, PhD, RD, Study Director — UAB, Department of Medicine; Ambika P Ashraf, MD, Study Director — Children's of Alabama, Pediatric Endocrinology
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Hanks LJ, Gutierrez OM, Ashraf AP, Casazza K. Bone Mineral Content as a Driver of Energy Expenditure in Prepubertal and Early Pubertal Boys. J Pediatr. 2015 Jun;166(6):1397-403. doi: 10.1016/j.jpeds.2015.02.054. Epub 2015 Apr 1. PMID 25841541